CLINICAL TRIAL: NCT01236846
Title: Determination of VDR Single Nucleotide Polymorphisms (SNPs ) and Their Rols in Efficacy of Vitamin D-fortified Yogurt Drink on the Metabolic-, Inflammatory - and Oxidative Stress Parameters in Type 2 Diabetic Patients
Brief Title: Vitamin D Receptor Polymorphisms and Efficacy of Vitamin D-Fortified Yogurt Drink in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tirang R. Neyestani (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Tirang R. Neyestani, associate professor, National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ABT-1236-RV
Record Dates: First submitted 2010-08-09; First posted 2010-11-09 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Vitamin D fortification; Yogurt Drink; Efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Plain Yogurt Drink (Placebo Comparator): Daily intake of unfortified yogurt drink(500 ml) for 12 weeks
  Interventions: Dietary Supplement: Plain Yogurt Drink
- VDR Genotype (aa) (Experimental): Daily intake of yogurt drink fortified (500 ml) with 1000IU vitamin D for 12 weeks
  Interventions: Dietary Supplement: Fortified Yogurt Drink
- VDR Genotype (AA) (Experimental): Daily intake of yogurt drink fortified (500 ml) with 1000 IU vitamin D for 12 weeks
  Interventions: Dietary Supplement: Fortified Yogurt Drink
- VDR genotype (Aa) (Experimental): Daily intake of yogurt drink fortified (500 ml) with 1000IU vitamin D for 12 weeks
  Interventions: Dietary Supplement: Fortified Yogurt Drink

INTERVENTIONS:
Dietary Supplement: Fortified Yogurt Drink — Daily intake of yogurt drink fortified (500 ml) with 1000IU vitamin D for 12 weeks
  Other Names: FYD
  Arms: VDR Genotype (AA); VDR Genotype (aa); VDR genotype (Aa)
Dietary Supplement: Plain Yogurt Drink — Daily intake of unfortified yogurt drink(500 ml)for 12 weeks
  Other Names: PYD
  Arms: Plain Yogurt Drink

SUMMARY:
Study is a 12-week Double blind,controlled experiments designed to examine the possible effects of vitamin D receptor gene polymorphisms on the metabolic, inflammatory and oxidative stress markers in type 2 diabetic patients to vitamin D-fortified yogurt drink intake.

DETAILED DESCRIPTION:
In a 12-week randomized controlled trial ( double-blind study), based on data on serum 25(OH)D changes from other studies (35), to achieve 1 standard deviation difference in circulating 25(OH)D with two-sided alpha of 0.05 and a beta of 0.2 after a 12-week intervention period, the sample size was calculated 40 individuals per treatment group. Considering 3 polymorphic variant groups and one control group which receives plain yogurt drink, 160 subjects are needed. Allowing for 10% attrition over 12 weeks of intervention, a total of 180 subjects are required. In treatment groups, all patients receive 500 ml per day of low-fat (1%) Yogurt Drink fortified with approximately 500IU of vitamin D3 . Control group receives 500 ml per day of plain (unfortified) Yogurt Drink. Metabolic, inflammatory and oxidative stress markers are evaluated at the beginning and in the end of the interventional period.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Informed consent
* BMI between 25 to 35 kg/m2
* Age: 30-45 years old
* Willingness to maintain current body weight for the duration of the study
* Willingness to maintain baseline lifestyle activities and routines for the duration of the study
* Willingness to avoid the use of all over-the-counter or prescription vitamins, dietary supplements, and herbal products during the study

Exclusion Criteria:

* History of cardiovascular , Gastrointestinal , Renal disease and any other endocrinological disorders
* Subjects receiving vitamin D or omega-3 supplement
* Pregnancy , or lactation within the study period
* Treatment with insulin
* Treatment for weight reduction
* Treatment for reducing serum lipids

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D | 3 months

SECONDARY OUTCOMES:
Glycemic control | 3 Months
Inflammatory markers | 3 Months
Oxidative stress markers | 3 Months
Lipid profiles | 3 Months
Blood pressure | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, Ph.D., Study Chair — National Nutrition & Food technology Research institute, P.O. Box 19395-4741; Abolghasem Djazayeri, Professor, Study Chair — Tehran University of Medical Sciences; Sakineh Shab-Bidar, M.Sc., Principal Investigator — Tehran University of Medical Sciences
Locations (3):
- Iran (3):
  - National Nutrition and Food Technology Research Institute, Tehran, Tehran Province
  - Tirang Neyestani, Tehran, Tehran Province
  - Tehran

REFERENCES:
- [Derived] Neyestani TR, Djazayery A, Shab-Bidar S, Eshraghian MR, Kalayi A, Shariatzadeh N, Khalaji N, Zahedirad M, Gharavi A, Houshiarrad A, Chamari M, Asadzadeh S. Vitamin D Receptor Fok-I polymorphism modulates diabetic host response to vitamin D intake: need for a nutrigenetic approach. Diabetes Care. 2013 Mar;36(3):550-6. doi: 10.2337/dc12-0919. Epub 2012 Nov 16. PMID 23160722
- [Derived] Shab-Bidar S, Neyestani TR, Djazayery A, Eshraghian MR, Houshiarrad A, Kalayi A, Shariatzadeh N, Khalaji N, Gharavi A. Improvement of vitamin D status resulted in amelioration of biomarkers of systemic inflammation in the subjects with type 2 diabetes. Diabetes Metab Res Rev. 2012 Jul;28(5):424-30. doi: 10.1002/dmrr.2290. Epub 2012 Feb 17. PMID 22344966
- [Derived] Shab-Bidar S, Neyestani TR, Djazayery A, Eshraghian MR, Houshiarrad A, Gharavi A, Kalayi A, Shariatzadeh N, Zahedirad M, Khalaji N, Haidari H. Regular consumption of vitamin D-fortified yogurt drink (Doogh) improved endothelial biomarkers in subjects with type 2 diabetes: a randomized double-blind clinical trial. BMC Med. 2011 Nov 24;9:125. doi: 10.1186/1741-7015-9-125. PMID 22114787
- [Derived] Shab-Bidar S, Neyestani TR, Djazayery A. Efficacy of vitamin D3-fortified-yogurt drink on anthropometric, metabolic, inflammatory and oxidative stress biomarkers according to vitamin D receptor gene polymorphisms in type 2 diabetic patients: a study protocol for a randomized controlled clinical trial. BMC Endocr Disord. 2011 Jun 22;11:12. doi: 10.1186/1472-6823-11-12. PMID 21696575